CLINICAL TRIAL: NCT04941664
Title: Minimum Effective Local Anesthetic Volume of 0.5% Levobupivacaine Required for Ultrasound Guided Superior Trunk Block for Shoulder Surgery
Brief Title: Minimum Effective Local Anesthetic Volume for Ultrasound Guided Superior Trunk Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC.2021.184-T
Record Dates: First submitted 2021-06-09; First posted 2021-06-28 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-05

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Superior Trunk nerve block
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Levobupivacaine

STUDY DESIGN:
Masking Description: Participants will be blinded to the amount of local anesthetic agent used. Outcome assessor assessing the outcomes will be blinded of the amount of local anaesthetic used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Levobupivacaine (Other): Superior trunk nerve block will be done under ultrasound guidance to patients scheduled for shoulder surgeries. Local anesthetic agent (0.5% levobupivacaine) 8ml will be injected at the superior trunk of the brachial plexus in order to produce surgical anesthesia or analgesia for shoulder surgeries.
  Interventions: Drug: 0.5% levobupivacaine

INTERVENTIONS:
Drug: 0.5% levobupivacaine — This study adopts a "Modified Narayana rule (MNR)", a sequential up-and-down pharmacodynamics method (UDM) to estimate the minimum effective local anesthetic volume of 90% (MELVA90) of cases of the aforementioned local anesthetic (LA), in order to produce the surgical anesthesia of the patients scheduled for shoulder surgeries. Based on the principal investigator's clinical experience, the initial volume of 8ml will be used. Depending on the success or failure of the superior trunk block, which is defined as the readiness for surgery at 30 minutes after the block, the volume for the next patient will be adjusted up or down by 2ml. The upper dose limit of the study to minimize the potential for local anesthetic systemic toxicity will be 16ml and the lower dose limit will be 4ml, which will be of no clinical importance.
  Other Names: Peripheral nerve block

SUMMARY:
The objective of this study is to identify the minimum effective dosage of a commonly used local anaesthetic drug "levobupivacaine" required to produce an effective ultrasound guided (USG) superior trunk block (STB) in at least 90% of patients for shoulder arthroscopic surgeries.

DETAILED DESCRIPTION:
Shoulder arthroscopic surgery is one of the most commonly performed procedures worldwide, and associated with significant postoperative pain. Currently, such surgery is performed either under general anaesthesia or under Interscalene brachial plexus block (ISBPB), which is a regional anaesthesia technique. However, ISBPB is associated with the highest incidence of hemi-diaphragmatic palsy of the operative side. Since majority of the innervation to the shoulder arises from or passes through the superior trunk of the brachial plexus, superior trunk block has been shown to have lesser impact on the phrenic nerve and it has been gaining popularity worldwide. Ultrasound is widely used for brachial plexus block and current evidence indicates that it is feasible to accurately identify majority of the main components of the brachial plexus above the clavicle, including the three trunks (superior, middle, and inferior trunks). However, there are no data describing an optimal volume of local anaesthetic for superior trunk block. The aim of this study is to identify the minimum effective dosage of a commonly used local anaesthetic drug "levobupivacaine" required to produce an effective ultrasound guided (USG) superior trunk block (STB) in at least 90% of patients for shoulder arthroscopic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III scheduled to undergo elective upper shoulder arthroscopic rotator cuff repair procedure

Exclusion Criteria:

* Patient refusal
* pregnancy
* skin infection at the site of block placement
* history of allergy to local anaesthetic drugs
* bleeding tendency or with evidence of coagulopathy
* pre-existing neurological deficit or neuromuscular disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes of sensory & motor blockade (Readiness for surgery) of the upper extremity | within 45 minutes after the block at 5 minutes interval
  The first exact timing (in minutes) [Readiness for surgery] that an Overall sensory score =<30 (NRS: 0-100; 100=normal sensation, 0=no sensation) using ice test and a motor grade =<1 (3 point scale: 2=no block, 1=paresis, 0=paralysis) in the nerves (C5 to C6) tested that are supplied by superior trunk of brachial plexus. Sensation to coldness (ice) will be tested at C5 - Lateral (radial) side of the antecubital fossa (just proximal to elbow crease); C6 - Thumb, dorsal surface, proximal phalanx. Motor block will be graded using a 3-points scale: 2=no block, 1=paresis and 0=paralysis, and will be test at C5 - elbow flexors and C6 - wrist extensors. "Block failure" will be defined as inability to achieve "readiness for surgery" at 30 minutes after the completion of the block.
Minimum effective volume (ml) of local anesthetic agent | after nerve block till end of surgery
  The lowest volume (in milliliters) of local anesthetic agent that can produce an effective superior trunk block for surgery. Effective superior trunk block is defined as an overall sensory score of NRS =<30 and a motor grade of =<1 during the assessment after the nerve block that can undergo surgery. Sensory assessment will be done by using ice (cold sensation) test in both dermatomes (C5, C6) and a motor grade of =<1 in both myotome (C5, C6) tested. Sensory block will be graded as 0 to 100 where 100 represents normal sensation and 0=no sensation to coldness (ice cube).

SECONDARY OUTCOMES:
Changes of motor blockade of the upper extremity | within 45 minutes after the block at 5 minutes interval
  Motor blockade will be graded using a 3-point scale: 2=no block, 1=paresis and 0=paralysis. Motor blockade of each individual nerve in the anaesthetized upper extremity will be evaluated by testing C5 - elbow flexors, C6 - Wrist extensors, C7 - Elbow extensors, C8 - Finger flexors to the middle finger, and T1 - small finger abductors. Onset of Motor block for each nerve will be defined as the time it took to achieve motor score =<1.
Changes of sensory block of the upper extremity | within 45 minutes after the block at 5 minutes interval
  Sensation to coldness (ice) will be test at C5- lateral (radial) side of the antecubital fossa (just proximal to elbow crease), C6 - Thumb, dorsal surface, proximal phalanx, C7 - middle finger, dorsal surface, proximal phalanx, C8 - Little finger, dorsal surface, proximal phalanx, and T1 - medial (ulnar) side of the antecubital) fossa, just proximal to the medial epicondyle of the humerus. Sensory block, defined as loss of sensation to cold (ice), will be graded using a numeric rating scale (NRS: 0-100, 100=normal sensation, 0=no sensation).
  Onset of sensory block for each nerve will be defined as the time that it took to achieve a sensory block score of NRS =<30.
Percentage changes of the Diaphragmatic function | Baseline (before block) and at 30 minutes after block
  Excursion of the ipsilateral hemidiaphragm will be measured by ultrasound machine in supine position via the anterior subcostal route. The movement of the diaphragm will be measured in centimetres. The range of diaphragmatic excursion will be recorded from the resting expiratory position to deep inspiration (sigh test) as will be the range of diaphragmatic movement from resting expiratory position when quickly inspiring through the nose (sniff test). The decrease in diaphragmatic excursion will be calculated as the difference (in %) in diaphragmatic excursion measured before and 30 minutes after superior trunk block (STB).
Changes of the Extensiveness of Diaphragmatic function | calculated after block
  After obtaining the percentage changes of the diaphragmatic function, if the reduction in diaphragmatic excursion of more than 75%, or no movement, or paradoxical movement will be considered as complete paresis. Reduction in diaphragmatic excursion of both sigh and sniff test between 25% and 75% will be considered as partial paresis and diaphragmatic excursion of less than 25% will be considered as 'no paresis'.
Block performance time | assess once before surgery
  The time taken from the start of the local anesthetic skin infiltration to the end of the injection of study drug for the nerve block.
Discomfort score | assess once before surgery
  the degree of discomfort during the nerve block (NRS: 0-100; 0= no discomfort, 100 = very uncomfortable)
Paresthesia | during the period of undergoing the nerve block
  Any incidence of paresthesia during the nerve block
Complications | during the nerve block till the end of surgery
  Any complications during and right after the nerve block directly related to local anesthetic toxicity, vascular or pleural puncture,intraneural injection with nerve swelling.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Anaesthesia & Intensive Care, Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No